CLINICAL TRIAL: NCT03769532
Title: MRD-guided Treatment With Pembrolizumab and Azacitidine in NPM1mut AML Patients With an Imminent Hematological Relapse
Brief Title: MRD-guided Treatment in NPM1mut AML Patients
Acronym: PEMAZA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Feasibility
Sponsor: Technische Universität Dresden (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TUD-PEMAZA-068
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; NPM1mut; molecular relapse; pembrolizumab; azacitidine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — pembrolizumab; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab + Azacitidine (Experimental): Pembrolizumab (IMP): 200 mg i.v. (fixed dose) / Azacitidine (SOC): 75 mg/m2 s.c.
  maximum duration of treatment: up to 24 weeks
  Interventions: Drug: Pembrolizumab; Drug: Azacitidine

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab (IMP): 200mg i.v. (fixed dose), every 3 weeks (Q3W), 8 doses
  Other Names: PEM; Keytruda®
Drug: Azacitidine — Azacitidine (SOC): 75 mg/m2 s.c., day 1-7 every 4 weeks (Q4W), 6 cycles
  Other Names: AZA; Vidaza®

SUMMARY:
Evaluation the safety and efficacy of Pembrolizumab (PEM) when administered in combination with standard Azacitidine (AZA) in nucleophosmin (NPM1) mutated AML patients with molecular relapse defined by the presence of measurable residual disease (MRD).

DETAILED DESCRIPTION:
Azacitidine is an effective and well established therapy in patients with acute myeloid leukemia (AML). In fact, in previous measurable residual disease (MRD) triggered studies, azacitidine allowed for a delay towards an overt hematological relapse in the majority of patients. However, the majority of patients ultimately relapsed even though they received multiple cycles of preemptive therapy. Hypomethylating agents (HMA) can enhance antitumor immune responses by upregulating tumor antigene expression, class 1 major histocompatibility complex, and co-stimulatory molecules, while concurrently dampening this antitumor effect by upregulating expression of checkpoint receptors or ligands, including programmed cell death protein 1 (PD-1), programmed cell death ligand 1 (PD-L1), and cytotoxic T-lymphocyte-associated protein 4 (CTLA-4). Upregulation of these immune checkpoint molecules might be a mechanism of resistance to hypomethylating drugs. It has been shown that PD-L1 Messenger ribonucleic acid (mRNA) is up-regulated acute myeloid leukemia cluster of differentiation 34 (CD34+) cells and importantly, patients resistant to treatment with hypomethylating agents such as azacitidine have an up-regulated expression compared to responding patients. In addition, it is known that PD-1 promoter demethylation correlates with a higher PD-1 expression and a worse response rate to hypomethylating agents as well as a shorter overall survival. In this context it is of note that PD-1 promoter demethylation can be caused by hypomethylating agents and hence the mode of action of the drug itself could cause resistance to therapy in these patients. This might also explain why hypomethylating agents are not curative and can not eradicate early leukemic progenitor cells. The investigators, therefore, perform a phase II trial evaluating a combination therapy of pembrolizumab and azacitidine in nucleophosmin (NPM1) mutated AML patients with MRD and impending hematological relapse after conventional chemotherapy. This trial aims at improving response rates observed with single agent azacitidine within the studies NCT00422890 and NCT01462578.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥18 years
* Patients with NPM1mut AML in complete morphologic remission after conventional chemotherapy (anthracycline ± cytarabine based)
* Detectable measurable residual disease (MRD) indicating imminent hematological relapse (NPM1mut MRD ratio >1%, confirmed by central lab)
* Patients who are not eligible for immediate allogeneic hematopoietic stem cell transplantation
* Patients who are not eligible to undergo alternative intensive treatment
* Intended AZA therapy for molecular relapse
* Eastern cooperative oncology Group (ECOG) performance status of 0 or 1
* Demonstrate adequate organ function as defined by protocol, all labs should be performed within the screening period.
* Negative pregnancy test in women of childbearing potential (negative urine or serum pregnancy within 3 days prior to receiving study treatment). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential (Section 5.9.2) must be willing to use an adequate method of contraception as outlined in Section 5.9.2 - Contraception, for the course of the study through 120 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Male subjects with procreative capacity (Section 5.9.2) must agree to use an adequate method of contraception as outlined in Section 5.9.2- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

* Prior allogeneic hematopoietic stem cell transplantation
* Treatment with any investigational drug within 4 weeks to study therapy or less than 5 half-lives preceding the first dose of trial medication, whichever is longer.
* Anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or no recovering (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or no recovering (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Prior treatment with an anti-programmed cell death protein (anti PD-1, anti PD-L1 or anti PD-L2 agent).
* Known hypersensitivity to any of the drugs within this study, their constituents or to drugs with similar chemical structure.
* Receiving immunosuppressive therapy within 7 days prior to the first dose of trial medication.
* Known history of active Bacillus Tuberculosis (TB).
* Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
* Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Known history of, or any evidence of active, non-infectious pneumonitis.
* Liver cirrhosis or malignant liver tumor.
* Known severe congestive heart failure, incidence of clinically unstable cardiac or pulmonary disease.
* Active infection requiring systemic therapy.
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Known Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., Hepatitis C virus (HCV) RNA [qualitative] is detected).
* Live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Proportion of event-free patients | after 24 weeks of combination treatment (i.e. after up to 6 cycles of AZA for 7 days every 4 weeks and up to 8 PEM infusions every 3 weeks)
  Events are:
  * First hematological relapse after start of combined therapy
  * Death from any cause
  * AML-treatment other than Pembrolizumab and Azacitidine or hypomethylating agents only

SECONDARY OUTCOMES:
Overall survival (OS) | through study completion, an average of 1 year
  Overall survival is defined as the number of days between date of first visit (AZA) and date of death from any cause.
Proportion of event-free patients | after 12 weeks of combined therapy
  For this endpoint apply the same definitions as for the primary endpoint.
Treatment-related mortality | during 24 weeks of combined therapy
  Any death without preceding hematologic relapse is considered to be treatment related.
Course of MRD-burden measured as quantitative NPM1/Abelson murine leukemia viral oncogene homolog 1 (ABL) ratio | through study completion, an average of 1 year
  The NPM1/ABL-ratio will be log-transformed with base 10. With the log transformation a near normal distributed variable will be derived to be able to use parametric methods for analysis. Values below limit of detection (LOD) will be substituted by LOD/2 before log-transformation.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Moritz Middeke, MD, Principal Investigator — Technische Universität Dresden (TUD)
Locations (10):
- Germany (10):
  - Klinikum Chemnitz, Chemnitz
  - Universitätsklinikum Dresden, Dresden
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Leipzig, Leipzig
  - Kliniken Maria Hilf, Mönchengladbach
  - Klinikum r. d. I., München
  - Universitätsklinikum Münster, Münster
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Universitätsklinikum Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No